CLINICAL TRIAL: NCT00585169
Title: A Phase II Open-Label Multi-Center Trial of Memantine (Namenda(TM)) Treatment of Pathological Gambling
Brief Title: Memantine Treatment Study of Pathological Gambling
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Minnesota (Other); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Marc Potenza, Professor of Psychiatry, Child Study, and Neurobiology, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0705002703*; HIC 0705002703 (Other: Yale University)
Record Dates: First submitted 2007-12-25; First posted 2008-01-03 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-03

CONDITIONS: Pathological Gambling
Keywords: Pathological Gambling; Compulsive Gambling; Gambling Addiction; Gambling; Treatment; Memantine; Pharmacology
MeSH Terms: conditions — Gambling | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- memantine (Experimental): 10 to 30 mg/day memantine. The study consisted of 10 weeks of open-label memantine. All eligible study subjects were started at 10 mg/day for 2 weeks. The dose was increased to 20 mg/day after 2 weeks and then to 30 mg/day after 4 weeks unless remission of PG symptoms was attained at a lower dose.
  Interventions: Drug: Memantine Hydrochloride

INTERVENTIONS:
Drug: Memantine Hydrochloride — 10 mg/day for two weeks, dose increase to 20 mg at week 3, 30 mg at week 4 unless clinical improvement is achieved with a lower dose. Total treatment is 10 weeks.
  Other Names: Namenda

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of the drug memantine in individuals with pathological gambling (PG). Thirty subjects with DSM-IV PG will receive 10 weeks of open-label treatment with memantine. The hypothesis to be tested is that memantine will be effective and well tolerated in patients with PG. We hypothesize that memantine will reduce the severity of gambling symptoms and improve patients' overall functioning. This study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pathological Gambling using the clinician-administered Structured Clinical Interview for Pathological Gambling (SCI-PG) (Grant et al., 2004);
* Gambling behavior within 2 weeks prior to enrollment;
* For women, negative results on a urine pregnancy test and stable use of a medically accepted form of contraception.

Exclusion Criteria:

* Infrequent gambling (i.e. less than one time per week) that does not meet DSM-IV criteria for PG;
* Unstable medical illness or clinically significant abnormalities on laboratory tests, EKG, or physical examination at screen;
* History of seizures;
* Myocardial infarction within 6 months;
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
* A need for medication other than memantine with possible psychotropic effects or unfavorable interactions;
* Clinically significant suicidality;
* Current Axis I disorder determined by the SCID and SCID-compatible modules for impulse control disorders (Grant et al., 2005), except for nicotine dependence;
* Lifetime history of bipolar disorder type I or II, dementia, schizophrenia, or any psychotic disorder determined by SCID;
* Current or recent (past 3 months) DSM-IV substance abuse or dependence;
* Positive urine drug screen at screening;
* Initiation of psychotherapy or behavior therapy within 3 months prior to study baseline;
* Previous treatment with memantine;
* Treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc N. Potenza, M.D, Ph.D., Principal Investigator — Yale University; Jon E Grant, MD, JD, MPH, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota

REFERENCES:
- [Result] Grant JE, Chamberlain SR, Odlaug BL, Potenza MN, Kim SW. Memantine shows promise in reducing gambling severity and cognitive inflexibility in pathological gambling: a pilot study. Psychopharmacology (Berl). 2010 Dec;212(4):603-12. doi: 10.1007/s00213-010-1994-5. Epub 2010 Aug 19. PMID 20721537
- See also: Drug info available from FDA's Drugs@FDA web site — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm
- See also: Yale University School of Medicine — http://info.med.yale.edu/ysm/
- See also: University of Minnesota Impulse Control Disorders Clinic — http://www.impulsecontroldisorders.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women with a primary diagnosis of Pathological Gambling (PG) were recruited between April 2008 through February 2010
Pre-assignment Details: Twenty-eight of the 29 enrolled subjects completed the study with only one subject withdrawing due to time constraints
Groups:
- Memantine: 10 to 30 mg/day memantine
  Memantine Hydrochloride : 10 mg/day for two weeks, dose increase to 20 mg at week 3, 40 mg at week 5 unless clinical improvement is achieved with a lower dose. Total treatment is 10 weeks. Mean dose at study end was 23.4 ± 8.1 mg/day
Period: Overall Study
Arm/Group | Memantine
Started | 29
Completed | 28
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale Modified for Pathological Gambling (PG-YBOCS)
Description: The PGYBOCS is a reliable & valid, 10-item, clinician administered scale that rates gambling symptoms within the last 7 days. The first 5 questions assess urges and thoughts associated with pathological gambling, and the last 5 questions assess the behavioral component of the disorder. Scores of 0 through 4 are assigned each item according to the severity of the response (0 = least severe response or none, 4 = most severe response or extreme)with a score ranging from 0-40. Each set of questions (1-5 and 6-10) can be totaled separately for the component score (urges/thoughts and behavioral) as well as together for a total score. A score of 0 indicates no problems while increasing scores indicate increasing severity of problems with gambling. PG-YBOCS is used to measure changes across time. A decreasing score indicates a possible positive response to the intervention. Total score at baseline was compared with the study end to determine if the intervention was efficacious.
Time Frame: Baseline to study end point (10 weeks)
Population: All participants who completed at least one study visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 29
units on a scale
  Baseline | 21.8 (4.3)
  10 weeks | 8.9 (7.2)

ADVERSE EVENTS:
Arm/Group | Memantine 10mg | Memantine 20mg | Memantine 30mg
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/24 | 0/16
Other Adverse Events (participants affected / at risk) | 5/29 | 6/24 | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine 10mg (N=29) | Memantine 20mg (N=24) | Memantine 30mg (N=16)
Light-headed/dizzy (General disorders) | 2 | 4 | 2
Headache (General disorders) | 3 | 0 | 0
Lethargic or tired (General disorders) | 0 | 1 | 3
Decreased libido (General disorders) | 0 | 1 | 1
Nausea (General disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No